CLINICAL TRIAL: NCT05049941
Title: Blood Gases Versus Lactate Clearance as an Indicator of Initial Resuscitation in Septic Patients: Comparative Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahmed Hassanein Mohamed, assistant professor, Minia University
Other Study IDs: 6382021
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Sepsis Syndrome
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome | interventions — Blood Gas Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- group1: Group (1): veno-arterial carbon dioxide tension / arteriovenous oxygen content P(v-a)CO2/C(a-v)O2 ratio group.
  Interventions: Diagnostic Test: lactat and blood gases
- group 2: Group (2): Lactate clearance (LC) group; Lactate level was measured then LC rate was calculated by the equation [(lactate(T0)- lactate(T8))/lactate(T0)] × 100%.
  Interventions: Diagnostic Test: lactat and blood gases
- group 3: Group (3):
  veno-arterial carbon dioxide tension group; P(v-a)co2 difference
  Interventions: Diagnostic Test: lactat and blood gases

INTERVENTIONS:
Diagnostic Test: lactat and blood gases — observational

SUMMARY:
- This perspective blind randomized single center study was designed to assess central venous and arterial gases level including P(v-a)CO2/C(a-v)O2 ratio and P(v-a)CO2 difference against lactate clearance as an indicator of initial resuscitation in septic patients in intensive care unit and to evaluate the success of early resuscitation protocol .this continuation of our previous work we compared the ratio of P(v-a)CO2/C(a-v)O2 ratio against lactate clearance(8). Mortality in the ICU in the study groups will be recorded

DETAILED DESCRIPTION:
On ICU admission, Criteria of Systemic Inflammatory Response Criteria (SIRS) were evaluated including: abnormal white blood cell count >12,000/ μL or <4000/ μL, heart rate >90/min, respiratory rate >20/min or PaCO2 < 32 mmHg or abnormal body temperature >38.3 °C (100.4 °F) or <36 °C (96.8 °F). The quick Sequential Organ Failure assessment (qSOFA) score (10) measured at the bedside : altered level of consciousness (Glasgow Coma Scale score ≤ 13), Systolic blood pressure < 90 mmHg and respiratory rate ≥ 22 rpm. The Acute Physiology and Chronic Health Evaluation (APACHE II) score were collected (Knaus et al.,1985). Patients monitoring of heart rate, pulse oximetry, invasive arterial blood pressure for measurement of MAP, core temperature (UltraviewSL2700; Spacelaps, USA). and urine output. Laboratory investigations includes: complete blood count, C-reactive protein, liver and renal functions, coagulation profile, blood glucose, sodium and potassium level. All patients had jugular central venous catheter was inserted under ultrasound guidance, and the position confirmed by chest radiograph, then central venous pressure (CVP) was measured before starting the initial resuscitation (T0) ansd 8 hours after resuscitation (T8). From CVP line, blood sample analyzed by (SIEMENS RAPIDPoint® 500 blood gas machine). The following measurements were recorded at (T0) and at (T8): Central venous oxygen saturation (ScvO2), Central venous oxygen tension (Pvo2) and Central venous carbon dioxide tension (Pvco2). The central venous oxygen content (Cvo2) Cvo2 = (1.34 × Svo2 × Hb) + (0.003 × Pvo2) Radial arterial canula was inserted under ultrasound guidance to all patients and arterial blood gases (ABG) was analyzed at (T0) and (T8) to measure: arterial oxygen tension (Pao2), arterial oxygen content (Cao2), arterial carbon dioxide tension (Paco2), arterial oxygen saturation (Sao2.) and lactate level Cao2 = (1.34 × Sao2 × Hb) + (0.003 × Pao2) Resuscitation Patients were randomly assigned (by computer generated sequence) into three groups each consists of 40 patients: Group (1): veno-arterial carbon dioxide tension / arteriovenous oxygen content P(v-a)CO2/C(a-v)O2 ratio group; Group (2): Lactate clearance (LC) group; Lactate level was measured then LC rate was calculated by the equation [(lactate(T0)- lactate(T8))/lactate(T0)] × 100%.

Group (3):

veno-arterial carbon dioxide tension group; P(v-a)co2 difference Measurements were obtained at T0 (before the start of resuscitation) and at T8 (after 8 hours of the start of resuscitation), the three groups received the same initial resuscitation protocol according to Surviving Sepsis Campaign (9), the appropriate specimens were taken for aerobic and anaerobic culture, empirical broad-spectrum antibiotics was given, source of infection was controlled with removal of any old intravascular lines which may be the source of sepsis.

The early goals of resuscitation were to achieve the following: CVP of 8-12 cmH2O, MAP > 65 mm Hg, a urine output >0.5 mL/kg and Scvo2 of 70% or more, we started with 30 ml/kg crystalloids in the first 3 hours, then we guided by hemodynamic status, if not achieved, we were targeted by titrating vasopressors until MAP > 65 mmHg by using either norepinephrine (0.25 mcg /kg/min increasing every 15 min) or dobutamine (2.5 mcg/min every 15 min increased). The patients connected to mechanical ventilation if needed with appropriate settings, with minimal dose of sedation, blood glucose controlled and anticoagulant and Proton pump inhibitors were administrated as a prophylaxis, early enteral nutrition was initiated, if there was no contraindications Measured data

In group (1) we prepared this measures at T0 and T8:

* The arteriovenous oxygen content difference (C(a-v)O2) C(a-v)O2 = Cao2 - Cvo2
* The venoarterial CO2 tension difference (P(v-a)CO2) P(v-a)CO2 = Pvco2 - Paco2
* P(v-a)CO2/C(a-v)O2 ratio

  * (Pvco2 - Paco2)/(Cao2 - Cvo2)

ELIGIBILITY:
Inclusion Criteria:

adult critically ill patients admitted to the ICU in Minia University Hospital. Patients Ages was ≥ 18 and ≤ 65 years including both sexs, resuscitation started after fulfilling the diagnostic criteria of sepsis issued by Surviving Sepsis Campaign 2016

Exclusion Criteria:

* We excluded Patients with chronic organ failure (Cardiovascular, Respiratory, Liver, Neurological and Renal.)

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 120 adult critically ill patients admitted to the ICU in Minia University Hospital. Patients Ages was ≥ 18 and ≤ 65 years including both sexs, resuscitation started after fulfilling the diagnostic criteria of sepsis issued by Surviving Sepsis Campaign 2016
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2021-11-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
in septic patients in intensive care unit and to evaluate the success of early resuscitation protocol | 3-4 monthes
  success of early resuscitation

CONTACTS AND LOCATIONS:
Overall Officials: ahmed hassanein, MD, Principal Investigator — Minia University
Locations (1):
- Ahmed Hassanein, Minya, Egypt